CLINICAL TRIAL: NCT00501527
Title: Immunotherapy With Depigmented and Polymerized Allergen Extract of Phleum Pratense in Patients Suffering From Allergic Rhinoconjunctivitis and/or Asthma
Brief Title: Immunotherapy With Depigmented and Polymerized Allergen Extract of Phleum Pratense
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laboratorios Leti, S.L. (Industry)
Responsible Party: Mª José Gómez, Laboratorios LETI S.L.Unipersonal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-001437-18; 6078-PG-OSL-145 (Other: Sponsor Protocol number)
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2010-12

CONDITIONS: Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic; Asthma
Keywords: Allergoid; Depigmented; Polymerized; Allergen-extract; Rhinoconjunctivitis; Asthma
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Conjunctivitis, Allergic; Asthma | interventions — Immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A: Biological vaccine (Experimental): The first active arm will receive a dose that is 10x less than the dose of the other arm
  Interventions: Biological: Immunotherapy with modified extract of P. pratense pollen
- B: biological vaccine (Experimental): The first active arm will receive a dose that is 10x more than the dose of the other arm
  Interventions: Biological: Immunotherapy with modified extract of P. pratense pollen
- C (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Immunotherapy with modified extract of P. pratense pollen — Sublingual (2 drops daily)
  Arms: A: Biological vaccine; B: biological vaccine
Other: Placebo — Placebo 2 drops daily
  Arms: C

SUMMARY:
The objective of this trial is to evaluate the clinical effectiveness of the administration of a depigmented and polymerized allergen extract of Phleum pratense in the rhinoconjunctivitis and/or asthma of slight or moderate intensity, due to allergy to grass pollen.

DETAILED DESCRIPTION:
Immunotherapy is a specific treatment for allergic diseases. Unlike conventional pharmacological treatment, immunotherapy is the only treatment that could modify the natural course of allergic disease. This is a prospective double-blind placebo controlled study with three arms of treatment: placebo and two active (one of the active arms will receive a dose that is 10x the dose of the other arm).

ELIGIBILITY:
Inclusion Criteria:

* Positive clinical history of allergy to Phleum pratense
* Patients of both gender aged from 12 up to 50 years.
* Positive prick test to Phleum pratense allergen extracts
* Specific IgE to Phleum pratense
* Positive clinical history of allergic rhinoconjunctivitis and/or asthma
* Written informed consent.

Exclusion Criteria:

* Use of immunotherapy during the last four years.
* Any contraindication for the use of immunotherapy in accordance with European Allergy and Clinical Immunology Immunotherapy Subcommittee criteria:
* Treatment with ß-blockers
* Coexistence of immunopathological diseases (e.g. of the liver, kidney, the nervous system, thyroid gland, rheumatic diseases) in which autoimmune mechanisms play a role
* Patients suffering from immune deficiencies
* Patients with serious psychiatric / psychological disturbances
* In addition, the following was considered as exclusion criteria:
* Pregnant or/ in lactation patients
* Patients aspirin intolerance

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2007-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Symptom scores | 1 year

SECONDARY OUTCOMES:
Nasal provocation test | 1 year
Dose-response skin prick-test | 1 year
Asthma quality of life questionnaire (AQLQ)/Rhinoconjunctivitis quality of life questionnaire (RQLQ) | 1 year
Medication scores | 1 year
Visual scales | 1 year
"In vitro" immunological tests | 1 year
Record of adverse events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Félix Lorente, Prf. PhD, Principal Investigator
Locations (1):
- Hospital Clínico de Salamanca, Salamanca, Salamanca, Spain